CLINICAL TRIAL: NCT07262099
Title: Study of Effects of Dao-yin Exercise on the Patients With Breast Cancer Post Operation and Receiving Adjuvant Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Chien-Jung Lin, Principal Investigator and Attending Physician, Department of Traditional Chinese Medicine, Tri-Service General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TSGH-C106-020
Record Dates: First submitted 2025-11-22; First posted 2025-12-03 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shangshou Dao-yin Group (Experimental): Participants practiced Shangshou Dao-yin, a traditional mind-body exercise, for 20 minutes daily throughout the course of adjuvant chemotherapy. A standardized instructional video was provided to guide home or hospital practice.
  Interventions: Behavioral: Shangshou Dao-yin
- Control Group (No Intervention): Participants received standard medical care during chemotherapy without any structured exercise intervention.

INTERVENTIONS:
Behavioral: Shangshou Dao-yin — Participants practiced Shangshou Dao-yin, a traditional Daoist mind-body exercise consisting of eight techniques: Bouncing, Rotation, Swaying, Swinging, Wobble, Chopping, and Abdominal (diaphragmatic) Breathing. The exercise features gentle, rhythmic movements combined with natural breathing and mental focus, and requires no equipment or special space, making it suitable for patients undergoing chemotherapy. A standardized instructional video, provided on DVD and through online streaming (e.g., YouTube), was used to guide self-practice. Participants performed 20 minutes of Shangshou Dao-yin per day throughout the entire course of adjuvant chemotherapy, either at home or in the hospital.
  Arms: Shangshou Dao-yin Group

SUMMARY:
This is a retrospective registration of a study that evaluated whether a traditional Dao-yin (mind-body exercise), called Shangshou Dao-yin, could improve sleep quality, Chinese medicine body constitution, and quality of life in breast cancer patients receiving adjuvant chemotherapy.

A total of 327 postoperative breast cancer patients completed baseline questionnaires. Among them, 150 eligible participants entered the trial and were assigned to either a Dao-yin exercise group (72 participants) or a control group (78 participants) based on their preference. The exercise group practiced 20 minutes of Shangshou Dao-yin daily throughout chemotherapy, while the control group received standard care only. After withdrawals, 138 participants completed the final evaluation (66 in the Dao-yin group and 72 in the control group).

Sleep quality, body constitution (BCQ), quality of life (EORTC), and chemotherapy-related adverse effects were assessed during treatment and three weeks after chemotherapy completion. The findings may help determine whether Shangshou Dao-yin can reduce sleep disturbance and enhance well-being during cancer treatment.

DETAILED DESCRIPTION:
Breast cancer remains one of the most prevalent malignant diseases among women, and many patients receiving adjuvant chemotherapy experience sleep disturbance, emotional distress, fatigue, and impaired quality of life.

Shangshou Dao-yin is a traditional Dao-yin (mind-body exercise) consists of eight techniques: Bouncing, Rotation, Swaying, Swinging, Wobble, Chopping, and Abdominal (diaphragmatic) Breathing. The core principle of the Shangshou Dao-yin method is to stimulate the lower dantian, the body's source of vital energy. Dao-yin emphasizes mental focus, natural breathing, and smooth, continuous movements that follow the body's structure to harmonize internal energy flow. It requires no equipment and minimal space, making it particularly suitable for patients during chemotherapy.

This retrospective registration describes a study that evaluated whether Shangshou Dao-yin could improve sleep quality, Chinese medicine body constitution, and health-related quality of life in breast cancer patients undergoing adjuvant chemotherapy. The study was approved by the Institutional Review Board of Tri-Service General Hospital (TSGHIRB-1-105-05-045) and was conducted between January 2017 and October 2019.

A total of 327 postoperative breast cancer patients completed baseline questionnaires. Among them, 150 eligible participants entered the trial and were assigned, based on preference, to either a Shangshou Dao-yin group (n = 72) or a control group (n = 78). The Dao-yin group practiced 20 minutes of Shangshou Dao-yin daily throughout chemotherap. A standardized instructional video, provided on DVD and through online streaming (e.g., YouTube) in collaboration with the Taiwan Society of Health Promotion. The control group received standard care only. After withdrawals, 138 participants (66 Dao-yin, 72 control) completed the final evaluation.

Data collection included baseline characteristics (age, sex, height, weight, marital status, education level, smoking and alcohol history, medical history, family history, pregnancy and childbirth history, food or drug allergies, and comorbidities). Cancer-related variables included TNM stage, surgical method, tumor histology, differentiation, hormone receptor status, and HER2 expression. Chemotherapy-related information included regimen, dosage, treatment cycles, dose modifications, delays, and completion of planned cycles.

Multiple clinical assessments were performed. Sleep quality was measured using the Chinese version of the Pittsburgh Sleep Quality Index (PSQI). Chinese medicine body constitution was assessed using the 44-item Body Constitution Questionnaire (BCQ), which measures Yang-Xu, Yin-Xu, and Stasis constitutions. Health-related quality of life was evaluated using the EORTC QLQ-C30 and QLQ-BR23. Psychological status was measured using the Beck Anxiety Inventory (BAI) and Beck Depression Inventory-II (BDI-II). Laboratory monitoring included white blood cell count, granulocyte and lymphocyte percentages, platelet count, hemoglobin, liver and kidney function tests, and electrolytes.

Chemotherapy-related adverse effects were documented according to the Common Terminology Criteria for Adverse Events (CTCAE v4.0), including hematologic changes, infection, gastrointestinal symptoms (nausea, vomiting, diarrhea, abdominal bloating), mucositis, neuropathy, skin pigmentation, and insomnia. Medication use was recorded, including supportive drugs for chemotherapy side effects, chronic disease medications, and complementary therapies such as Chinese herbal medicine or special diets. Unscheduled outpatient visits, emergency department visits, hospitalizations, and physician-directed management of serious toxicities (dose reduction, treatment delay, or discontinuation) were also documented.

Assessments were performed before chemotherapy, at scheduled 4 time points during treatment, and three weeks after completion of chemotherapy. This study may help determine whether a traditional mind-body exercise can be feasibly implemented as a supportive care strategy for breast cancer patients undergoing chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed Stage I, II, or III breast cancer with surgical tumor removal followed by adjuvant chemotherapy.
2. Age ≥ 20 years.
3. Ability to walk independently without movement restrictions.
4. Able to communicate in Mandarin or Taiwanese.
5. Provided written informed consent.

Exclusion Criteria:

1. Regularly practicing Tai Chi or other mind-body exercises at the time of enrollment.
2. Pre-existing chronic illnesses or symptoms that may interfere with evaluation of chemotherapy-related side effects (e.g., chronic diarrhea, neuropathy, heart failure, thromboembolic disease, chronic pulmonary or renal disease, alopecia).
3. Pregnancy.
4. Severe psychiatric illness (e.g., schizophrenia, major depressive disorder).

Ages: 20 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-01-13 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2019-11-08 (Actual)

PRIMARY OUTCOMES:
Change in Health-Related Quality of Life (EORTC Quality of Life Questionnaire-Core 30; QLQ-C30) | Baseline to 3 weeks after completion of chemotherapy
  Quality of life was assessed using the EORTC Quality of Life Questionnaire-Core 30 (QLQ-C30). Scores were transformed to 0-100 scales, with higher functional scores indicating better functioning and higher symptom scores indicating worse symptoms.
  Score Range: 0-100 Directionality: Higher = better (function scales); Higher = worse (symptom scales)
Change in Breast Cancer-Specific Quality of Life (EORTC Breast Cancer-Specific Quality of Life Questionnaire; QLQ-BR23) | Baseline to 3 weeks after completion of chemotherapy
  Breast cancer-specific quality of life was measured using the EORTC Breast Cancer-Specific Quality of Life Questionnaire (QLQ-BR23). All subscales were transformed to 0-100 scales, with higher functional scores indicating better functioning and higher symptom scores indicating worse symptoms.
  Score Range: 0-100 Directionality: Higher = better (function scales); Higher = worse (symptom scales)

SECONDARY OUTCOMES:
Change in Body Constitution (Body Constitution Questionnaire; BCQ) | Baseline to 3 weeks after completion of chemotherapy
  Body constitution was assessed using the Body Constitution Questionnaire (BCQ), a 44-item instrument scored on a 1-5 Likert scale evaluating Yang-Xu, Yin-Xu, and Stasis constitutions. Higher scores indicate greater deviation from a balanced (neutral) constitution.
  Score Range: 44-220 (total possible score range across 44 items scored 1-5) Directionality: Higher = worse (greater imbalance)
Chemotherapy-related Adverse Events (CTCAE v4.0) | Baseline to 3 weeks after completion of chemotherapy
  Chemotherapy toxicities were documented according to the Common Terminology Criteria for Adverse Events (CTCAE v4.0), including hematologic changes, gastrointestinal symptoms, mucositis, neuropathy, skin reactions, and infection.

OTHER OUTCOMES:
Sleep Quality (Pittsburgh Sleep Quality Index; PSQI) | Baseline to 3 weeks after completion of chemotherapy
  Sleep quality was assessed using the Pittsburgh Sleep Quality Index (PSQI), a 19-item questionnaire with a score range of 0 to 21, where higher scores indicate poorer sleep quality.
Anxiety (Beck Anxiety Inventory; BAI) | Baseline
  Anxiety was measured using the Beck Anxiety Inventory (BAI), a 21-item scale with a score range of 0 to 63, where higher scores indicate more severe anxiety symptoms.
Beck Depression Inventory-II; BDI-II | Baseline
  Depression was assessed using the Beck Depression Inventory-II (BDI-II), a 21-item instrument with a score range of 0 to 63, where higher scores indicate more severe depressive symptoms.
Hematologic and Biochemical Laboratory Parameters | Baseline to 3 weeks after completion of chemotherapy.
  Hematologic parameters include white blood cell count, granulocyte percentage, lymphocyte percentage, platelet count, and hemoglobin level.
  Biochemical parameters include liver function tests, renal function tests, electrolyte levels, and tumor markers.
  These laboratory values were collected as part of protocol-specified assessments.

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-Service General Hospital, Taipei, Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No